CLINICAL TRIAL: NCT03647111
Title: A Real World Study to Evaluate the Efficacy and Safety of First Line Crizotinib in ALK Rearranged Advanced Non Squamous Non-small Cell Lung Cancer
Brief Title: Real World Study of First Line Crizotinib for ALK Rearranged Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Other Study IDs: RECURE
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; ALK rearranged; Crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohorts 1
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib 250mg po bid

SUMMARY:
This study aims to explore the efficacy and safety of Crizotinib as a first-line therapy for advanced non-squamous non-small cell lung cancer with ALK-positive mutations in the real world.

DETAILED DESCRIPTION:
According to the study of P11014 and P1029, Crizotinib is a first-line therapy for advanced non squamous non small cell lung cancer with positive ALK rearrangement.This study aims to explore the efficacy and safety of clozotinib as a first-line therapy for advanced non-squamous non-small cell lung cancer with ALK-positive mutations in the real world. Among them, ALK positive was based on NGS test results, exploring the new drug resistance mechanism of ALK under clozotinib treatment mode and consistency between plasma and tissue detection driving genes, and finally assessing the role of plasma dynamic detection driving gene mutation spectrum in predicting disease progression risk. A retrospective study of 120 patients with advanced NSCLC using clozotinib ALK positive mutation was conducted to observe the efficacy and safety of clozotinib regimen in the real world.

ELIGIBILITY:
Inclusion Criteria:

* ≥18，Pathologically proven ALK positive mutation in advanced non squamous non small cell lung cancer
* ALK rearrangement detection method is NGS and Ventana
* Primary treatment of first diagnosis
* The treatment was Crizotinib 250mg po bid Exclusion Criteria
* Patients received antitumor treatment before
* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who diagnosed ALK positive mutation in advanced non squamous non small cell lung cancer treated by Crizotinib.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Approximately 1 years
  Progression free survival

SECONDARY OUTCOMES:
OS | Approximately 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhou Y, Song L, Xu Q, Zeng L, Jiang W, Yang N, Zhang Y. Investigation on the survival implications of PD-L1 expression status in ALK- rearranged advanced non-small cell lung cancer treated with first-line crizotinib. Lung Cancer. 2022 May;167:58-64. doi: 10.1016/j.lungcan.2022.04.002. Epub 2022 Apr 6. PMID 35405360
- [Derived] Zhang Y, Zeng L, Zhou C, Li Y, Wu L, Xia C, Jiang W, Hu Y, Liao D, Xiao L, Liu L, Yang H, Xiong Y, Guan R, Lizaso A, Mansfield AS, Yang N. Detection of Nonreciprocal/Reciprocal ALK Translocation as Poor Predictive Marker in Patients With First-Line Crizotinib-Treated ALK-Rearranged NSCLC. J Thorac Oncol. 2020 Jun;15(6):1027-1036. doi: 10.1016/j.jtho.2020.02.007. Epub 2020 Feb 27. PMID 32112982